CLINICAL TRIAL: NCT03652376
Title: Impact of Benralizumab Treatment on Circulating Dendritic Cells in Patients With Eosinophilic Asthma
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Rostock (Other)
Responsible Party: Principal Investigator, Marek Lommatzsch, Prof. Dr. Marek Lommatzsch, University of Rostock
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Rostock-Benralizumab-2018-1
Record Dates: First submitted 2018-08-26; First posted 2018-08-29 (Actual); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Severe Eosinophilic Asthma
MeSH Terms: conditions — Pulmonary Eosinophilia | interventions — benralizumab

STUDY DESIGN:
Intervention Model Description: Patients with severe eosinophilic asthma (n=20) will be treated with benralizumab 3 times every 4 weeks, and the effect of this treatment on dendritic cell concentrations and dendritic cell characteristics will be investigated 4 weeks after the last benralizumab dose and after a follow-up of 3 months. There will be a separate control group of subjects (not a treatment or placebo arm) without asthma not treated with benralizumab (to study dendritic cell concentrations and dendritic cell characteristics in patients without asthma and without benralizumab treatment).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Benralizumab (Experimental): Patients will be treated with Benralizumab 30 mg s.c. every 4 weeks (three times).
  Interventions: Drug: Benralizumab

INTERVENTIONS:
Drug: Benralizumab — Treatment with Benralizumab 30 mg s.c. every 4 weeks (three times)

SUMMARY:
This study investigates the effect of removing eosinophils from peripheral blood (using treatment with Benralizumab, which is approved for the treatment of severe eosoniphilic asthma) on circulating dendritic cells in patients with severe eosinophilic asthma.

DETAILED DESCRIPTION:
Phase III clinical trials demonstrated that benralizumab treatment results in a significant decrease in exacerbations and a significant increase in lung function and quality of life in patients with severe eosinophilic asthma. However, the precise underlying mechanisms leading to this clinical benefit of benralizumab treatment are not completely understood. Dendritic cells are key regulators of the adaptive and innate immune system. There is evidence that eosinophils have a direct influence on the function of dendritic cells. In addition, there are multiple indirect interactions between eosinophils and dendritic cells in asthma. However, there is currently no information on the impact of benralizumab treatment and a complete removal of circulating eosinophils on the number and phenotype of human dendritic cells. Benralizumab is chosen for this study because it is the only anti-IL-5 biologic which results in a complete removal of eosinophils from peripheral blood.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 75 years
2. Patients with severe eosinophilic asthma inadequately controlled despite high-dose inhaled corticosteroids plus long-acting β-agonists.
3. Documented reversibility of airway obstruction (FEV1 increase ≥ 200 ml and ≥ 15 % after inhalation of a short-acting beta agonist) or bronchial hyperresponsiveness to methacholine or histamine
4. Documented concentration of blood eosinophils ≥ 300 / µl blood on the day of study inclusion or in the previous 4 weeks before study inclusion
5. Documented current treatment with high daily doses of ICS plus at least one other asthma controller for at least 3 months at Visit 1.
6. Disease history: asthma exacerbations while on ICS plus another controller.
7. ACQ-6 score ≥ 1.5 at Visit 1.
8. Weight of ≥ 40 kg.
9. Screening pre-bronchodilator (pre-BD) FEV1 of < 80% predicted
10. Women of childbearing potential (WOCBP)(Definition: WOCBP are those women who have not been surgically sterilized or have not been free from menses for > 2 years) and male study participants have to use adequate contraception methods.

Exclusion Criteria:

1. Smoking history of > 10 Pack years
2. Current smoking
3. Presence of other chronic pulmonary diseases including COPD
4. Presence of other chronic inflammatory diseases
5. Treatment with any systemic immunosuppressive drug including prednisolone or biologics
6. Current pregnancy, breast feeding
7. Known helminth infections
8. Acute upper or lower respiratory infections within 30 days prior to the date informed consent is obtained or during the screening/run-in period.
9. Any disorder, including, but not limited to, cardiovascular, gastrontestinal, hepatic, renal, neurological, musculosceletal, infectious, endocrine, metabolic, hematological, psychiatric, or major physical impairment that is not stable in the opinion of the Investigator and could:

   * affect the safety of the patient throughout the study
   * influence the findings of the studies or their interpretations
   * impede the patient´s ability to complete the entire duration of study
10. Hypersensitivity to the active substance or to any of the excipients listed in section 6.1 of the SmPC.
11. A helminth parasitic infection diagnosed within 24 weeks prior to the date informed consent is obtained that has not been treated with, or has failed to respond to, standard of care therapy.
12. Any clinically significant abnormal findings in physical examination, vital signs, hematology, or clinical chemistry during screening period, which in the opinion of the investigator may put the patient at risk of his/her participation in the study, or may influence the results of the study, or the patient´s ability to complete entire duration of the study.
13. Any clinically significant cardiac disease or any electrocardiogram (ECG) abnormality which in the opinion of the Investigator may put the the patient at risk or interfere with study assessments.
14. A history of known immunodeficiency disorder including a positive human immunodeciency virus (HIV) test.
15. Current malignancy, or history of malignancy, except for: Patients who have had non-melanoma skin cancer or in situ carcinoma of the cervix are eligible provided that the patient is in remission and curative therapy was completed at least 12 months prior to the date informed consent is obtained. Patients who have had other malignancies are eligible provided that the patient is in remission and curative therapy was completed at least 5 years prior to the date informed consent is obtained.
16. Concurrent biologics for asthma are not allowed except for stable allergen immunotherapy (defined as a stable dose and regimen at the time of Visit 1). Acceptable washout periods or other asthma biologics:

    * Other eosinophil lowering products indicated for asthma (including reslizumab or mepolizumab): at least 4 months.
    * Prior omalizumab use: 1 month.
17. Any immunosuppressant systemic medication (including systemic glucocorticoids) or treatment with antibodies targeting the immune system.
18. Receipt of any investigational medication as part of a research study within approximately 5 half-lives prior to randomization
19. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) level > 3 times of the upper limit of normal (ULN) confirmed during screening period.
20. Receipt of immunoglobulin or blood products within 30 days prior to the date informed consent is obtained.
21. Receipt of live attenuated vaccines 30 days prior to the date of randomization; other types of vaccines are allowed.
22. Planned surgical procedures during the conduct of the study.
23. Concurrent enrolment in another interventional or post-authorization safety study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-09-01 (Estimated); Primary Completion 2019-05-01 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Dendritic cell concentrations and phenotypes | 5 months
  Dendritic cell concentrations and phenotypes

SECONDARY OUTCOMES:
T-cell concentrations and phenotypes | 5 months
  T-cell concentrations and phenotypes

CONTACTS AND LOCATIONS:
Overall Officials: Marek Lommatzsch, MD, Principal Investigator — University of Rostock
Locations (1):
- University of Rostock, Rostock, Mecklenburg-Vorpommern, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lommatzsch M, Marchewski H, Schwefel G, Stoll P, Virchow JC, Bratke K. Benralizumab strongly reduces blood basophils in severe eosinophilic asthma. Clin Exp Allergy. 2020 Nov;50(11):1267-1269. doi: 10.1111/cea.13720. Epub 2020 Aug 26. No abstract available. PMID 32762056